CLINICAL TRIAL: NCT00773539
Title: Safety and Efficacy of Transvenous Pulmonary Isolation for the Treatment of Atrial Fibrillation: A Prospective Randomized Study Comparing Radiofrequency Energy With Cryoenergy
Brief Title: A Prospective Randomized Study Comparing Radiofrequency Energy With Cryoenergy
Acronym: CRYO-RF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Collaborators: CryoCath Technologies Inc. (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Thomas Arentz, Herz-Zentrum Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRYO-BAD-KROZ
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Atrial Fibrillation Ablation
Keywords: atrial fibrillation; pulmonary veins; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Procedure: PVI using an open irrigated tip catheter
- 2 (Active Comparator)
  Interventions: Procedure: PVI using a closed irrigated tip catheter
- 3 (Active Comparator)
  Interventions: Procedure: PVI using a cryoballoon

INTERVENTIONS:
Procedure: PVI using an open irrigated tip catheter — transseptal PVI using thermocooled ablation catheter (Biosense) with confirmation of conduction block
  Arms: 1
Procedure: PVI using a closed irrigated tip catheter — transseptal PVI using the CHILLI II catheter from BOSTON with confirmation of conduction block
  Arms: 2
Procedure: PVI using a cryoballoon — transseptal PVI using the cryoballoon from CRYOCATH
  Arms: 3

SUMMARY:
Transvenous pulmonary vein (PV) isolation using radiofrequency energy is an effective treatment for atrial fibrillation (1-4). However, rare but potentially life threatening complications such as thromboembolism (5), PV stenosis (5-10), left atrium-oesophageal fistula (11) and inflammatory syndromes (12) have been described. In preliminary studies an alternate approach using cryoenergy induces less endothelial disruption/ thrombus formation (13), preserves the extra cellular matrix and creates lesions with well-delineated border zones (14). Therefore, cryoenergy seems to be the ideal form of energy to safely perform PV isolation.

We therefore hypothesise that in the setting of PV isolation for the treatment of atrial fibrillation (AF) cryoenergy is less traumatic and therefore reduces systemic inflammatory responses compared to radiofrequency energy.

78 patients presenting with symptomatic intermittent or persistent AF will be randomised to PV isolation with either radiofrequency (26 patients open irrigated tip, 26 patients closed irrigated tip) or cryoenergy (26 patients with cryoballoon). Systemic markers of cell damage and inflammatory response (t-troponin, CK, CK-MB, vWF, PAI-1, micro particles, platelet activation/overall function, CRP, IL-6, IL-8, IL-10, TNF alpha, procalcitonin) will be monitored before, during and 48h after the procedure. Further endpoints include time to PV-isolation and procedure related complications. Six month clinical follow-up will focus on freedom from AF and cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Symptomatic drug refractory (more than 2 antiarrhythmic drugs) paroxysmal or persistent AF
* Documentation of AF on 12 lead ECG and/ or Holter
* Left atrium of less than 55 mm
* Informed consent signed by the patient

Exclusion Criteria:

* Previous Ablation or operation for AF
* Contra-indication for heart catheterisation
* Cardioversion for AF during the 2 weeks before the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-02 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Changes of platelet function (number of patients with an increase of more than 100% in platelets positive for either P-selectin or activated GP IIb/IIIa) | before, at the end of intervention, 6, 24 and 48 hours later.

SECONDARY OUTCOMES:
Parameters of inflammation and tissue damage, the time to achieve PV-Isolation, freedom from AF. | before, during and 6 months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Herz-Zentrum, Bad Krozingen, Germany

REFERENCES:
- [Derived] Jesel L, Arentz T, Herrera-Siklody C, Trenk D, Zobairi F, Abbas M, Weber R, Minners J, Toti F, Morel O. Do atrial differences in endothelial damage, leukocyte and platelet activation, or tissue factor activity contribute to chamber-specific thrombogenic status in patients with atrial fibrillation? J Cardiovasc Electrophysiol. 2014 Mar;25(3):266-70. doi: 10.1111/jce.12312. Epub 2013 Nov 22. PMID 24172190
- [Derived] Herrera Siklody C, Arentz T, Minners J, Jesel L, Stratz C, Valina CM, Weber R, Kalusche D, Toti F, Morel O, Trenk D. Cellular damage, platelet activation, and inflammatory response after pulmonary vein isolation: a randomized study comparing radiofrequency ablation with cryoablation. Heart Rhythm. 2012 Feb;9(2):189-96. doi: 10.1016/j.hrthm.2011.09.017. Epub 2011 Sep 13. PMID 21920484